CLINICAL TRIAL: NCT00886327
Title: Detection of Postoperative Recurrence of Crohn's Disease by Colonic Capsule-Endoscopy
Brief Title: Detecting Postoperative Recurrence in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Joerg Albert, MD, Medizinische Klinik 1, Klinikum der J. W. Goethe-Universität Frankfurt am Main
Other Study IDs: JWGUHMED1-001
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2009-04

CONDITIONS: Crohn's Disease
Keywords: Colonic capsule endoscopy; Crohn's disease; Capsule endoscopy
MeSH Terms: conditions — Crohn Disease | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Postoperative patients: Patients with CD who recently underwent bowel resection
  Interventions: Procedure: Colonic capsule endoscopy

INTERVENTIONS:
Procedure: Colonic capsule endoscopy

SUMMARY:
Up to ¾ of patients who have been diagnosed with Crohn's disease (CD) will have to undergo bowel resection during their lifetime despite modern medical therapies. Unfortunately, disease recurrence is common and endoscopic detection of recurring inflammation precedes clinical relapse. Endoscopic investigation is therefore recommended to manage these patients.

This multi center, prospective study compares the conventional endoscopic method, ileo-colonoscopy to a new technique, i.e., colonic capsule endoscopy (CCE). CCE enables investigation of the small bowel and the large intestines by using a double-sided video camera with about 10 hours acquisition time.

This study aims to evaluate the performance of CCE to detect postoperative recurrence of CD and detection rate of colonic and anastomotic recurrence is compared to ileo-colonoscopy. Proximal (small bowel) lesions are additionally recorded and impact on clinical management of the findings is accounted for. Moreover, safety aspects and influence of the findings on progress of the disease are monitored. All consecutive patients who are operated for CD in any of the participating study centers are eligible. Included are patients with segmental small bowel, ileocecal or segmental colonic resection.

In some cases capsule retention has been reported at an average of 2-3% with CD patients at elevated risk. Therefore, patency capsule is performed before application of the video CCE to exclude bowel obstruction.

Sample size estimation results in n = 70, requiring each 140 capsule endoscopes and 140 patency capsules for performance of postoperative screening (ca 4-8 weeks postoperatively) and detection of postoperative recurrence (ca 4-8 months postoperatively).

ELIGIBILITY:
Inclusion Criteria:

* Segmental bowel resection for Crohn's disease

  * Ileocecal resection
  * Small bowel resection
  * Segmental colonic resection
* Informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Intestinal obstruction as suspected by anamnesis or clinical/technical investigation
* Dysphagia or ileus
* Non-passage of the intact 'Agile Patency Capsule' within 72 hours
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who are operated for CD in any of the participating study centers are eligible. Included are patients with segmental small bowel, ileocecal or segmental colonic resection. All patients have to give written informed consent before participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Detection of postoperative recurrence of CD

SECONDARY OUTCOMES:
Therapeutic intervention due to detection of recurrent CD
Detection of small bowel lesions by CCE
Rate of bowel stenosis as detected by PC
Side effect of CCE and/or colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Joerg G Albert, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (4):
- Germany (4):
  - Klinikum der JW Goethe Universität Frankfurt, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklnikum Leipzig, Leipzig
  - Klinikum der Universität München - Campus Grosshadern, München